CLINICAL TRIAL: NCT06549712
Title: The Fondazione Genomic SARS-CoV-2 Study
Brief Title: The Fondazione Genomic SARS-CoV-2 Study COVID-19
Acronym: FOGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Valenti:, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FOGS
Record Dates: First submitted 2024-03-07; First posted 2024-08-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-08

CONDITIONS: COVID-19; Genetic Predisposition
MeSH Terms: conditions — COVID-19; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- identify the main common genetic determinants (Experimental): The purpose of the entire project is to identify genetic determinants of the predisposition to develop respiratory failure in persons infected by SARS-CoV-2; knowledge of these factors may educate the biological understanding of the development of severe lung disease in SARS-CoV-2 infection. Such an understanding may inform treatment trials of potential utility towards more effective management of this patient group. A polygenic risk score may also be useful in identifying high/low risk patients, e.g. amongst health-care providers and vulnerable individuals with significant comorbidities.
  Interventions: Genetic: genetic determinants to develop respiratory failure

INTERVENTIONS:
Genetic: genetic determinants to develop respiratory failure — To identify the main common genetic determinants of severe COVID-19 by conducting a GWAS: in first phase we will compare SARS-CoV-2 positive patients with severe lung affection to healthy controls from the same geographic area, in order to provide initial data informing the research in the field in a timely fashion. This will be conducted in close collaboration with the University of Kiel COVID-19 genomic initiative. Later on, we will proceed to assess objectives 1 and 2 in the full cohort, including also infected controls who did not developed clinically significant symptoms
Genetic: genetic determinants to develop respiratory failure — To provide extensive genetic characterization of all patients managed at the Fondazione in order to facilitate other groups working on specific projects (e.g. on candidate genes such as SERPINA1 and ACE2 by the Intensive Care and Cardiology Units and other that may emerge from upcoming projects), in a large population and in a very timely fashion, and without incurring in any additional expenses for the Fondazione research network, and coordinate research efforts.
Genetic: genetic determinants to develop respiratory failure — To provide a coordination to manage the collaboration with other research consortia in the field, e.g. the "An anonymized GWAS to urgently query host genetic predisposition to severe COVID-19 (SARS-CoV-2 infection) lung disease, and the COVID-19 Host Genetic Initiative (https://www.covid19hg.org). Indeed, collaboration among large networks analyzing several thousand cases will be ultimately necessary to clarify the genetic basis of COVID-19 susceptibility, and large collaborative networks are essential instruments for conducting human genetic research.

SUMMARY:
Genetic association at the genomic level (genomewide association study - GWAS), requencing by NGS (whole exome sequencing) and gene expression studies to identify the main ones hereditary genetic determinants of predisposition to the development of SARS (symptomatic pathology associated with development of insufficiency respiratory disease of any degree) in Italian subjects affected by SARSCoV-2.

DETAILED DESCRIPTION:
Lombardy region in Northern Italy is now in the midst of an outbreak of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus that causes coronavirus disease 2019 (COVID-19) . The COVID-19 epidemic situation needs little introduction and represent a global world-wide emergency with mortality rates rapidly increasing in Europe and the US. Evidence is accumulating that the majority of individuals infected by SARS-CoV-2 are asymptomatic and the major source of viral spread 3, and that a considerable fraction of these has active viral replication 4,5. Furthermore, disease behavior is variable, with the majority of patients experiencing only mild symptoms or no symptoms at all. Some patients develop severe pulmonary affection, with aggressive and extensive inflammatory destruction of lung parenchyma and associated inflammatory responses and superinfections, driving large fractions of the COVID-19 related mortality. What exactly drives this development of severe lung disease remains unknown, but old age, obesity, diabetes and other co-morbidities increase the risk, while the role played by specific medications is still uncertain. Variation in virus genetics and patient immunology are also likely involved. As to the latter point, the investigators hypothesize that host genetics may play a role in determining development of severe lung disease in SARS-CoV-2 infection. Genome-wide association studies (GWAS) have been applied to decipher the genetic predisposition in thousands of disease traits since the study design was invented in 2005. The genetic signals detected vary from very strong effects that can be detected in a few hundred individuals, to very weak effects requiring cohorts of tens of thousands for detection. By 2020, the study design is now a robust, off-the-shelf, easyto-perform industry-standard screening tool for genetic predisposition, even available through "consumer genetics" online-based companies. The study design is simple: testing for genetic variants throughout the genome (single nucleotide polymorphisms, SNPs) using SNP microarrays, comparing their frequencies in patients versus controls (or across other variables). For inflammatory phenotypes in particular, GWAS has proven an efficient tool, delineating hundreds of susceptibility loci in many conditions, some of which has provided novel and surprising disease insights. GWAS serve two purposes. Most importantly they allow to determine biological factors involved in disease development, thus potentially guiding drug development and therapy. This would be particularly relevant during the current COVID-19 emergency, when hundreds of trials have begun and there is an urgent need to prioritize well-conducted collaborative studies based on robust pathophysiological data. Secondly, and increasingly popular, they allow for the calculation of a "polygenic risk score" to predict disease development. Both aspects appear crucial to clarify for COVID-19 lung disease: (a) are there genetic signatures suggesting which biological mechanisms are involved that may suggest relevant therapeutic approaches, and (b) can we predict those at risk (or those with very low risk)?

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 inclusion criteria:

* SARS-CoV-2 positive patients (no age limit) with severe pulmonary compromise, hospitalized with failure respiratory that requires support of any kind
* Signature of informed consent

Cohort 2 inclusion criteria:

* Blood donors (18-70 years old) who donated between 24/02/2020 and 31/12/2021
* exposure to the SARS-CoV-2 virus confirmed by viremia positive and presence of IgG/IgM
* Signature of informed consent

Cohort 3 inclusion criteria:

Healthy controls available from previous studies (n=5,000, ages 14-80 years), whose data are already available for genetic association analyses within the Kiel University database.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
SNPs as identified by GWAS | up to 36 months
  We will measure the differences in genetic background between patients with severe SARS-CoV-2 infection and healthy controls from the same geographical area, and identify the genetic differences between patients with severe SARSCoV infection2 and those with mild or moderate infection.

SECONDARY OUTCOMES:
rare genetic variants identified by Whole Exome sequencing (WES) | up to 36 months
  Examine the possible role of rare genetic variants in determining severe COVID-19 susceptibility in individuals who have developed severe respiratory failure despite lack of comorbidity and risk factors.
  Deidentified DNA samples will be sequenced to assess the genetic risk profile at the genomic level. In addition, the frequency distributions of common genetic variants will be compared between donors who have eliminated infection without developing severe symptoms and patients hospitalized for respiratory failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT06549712/Prot_SAP_000.pdf